CLINICAL TRIAL: NCT00706082
Title: A Two-stage Prospective Observational Cohort Study in Scleroderma Patients to Evaluate Screening Tests and the Incidence of Pulmonary Arterial Hypertension and Pulmonary Hypertension
Brief Title: Early, Simple and Reliable Detection of Pulmonary Arterial Hypertension (PAH) in Systemic Sclerosis (SSc)
Acronym: DETECT
Status: Terminated | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-052-510
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Systemic Sclerosis; Pulmonary Arterial Hypertension; Pulmonary Hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be stored at a central laboratory for at least two additional years after official study termination.
Oversight: Data Monitoring Committee: No

SUMMARY:
A two-stage prospective observational cohort study in scleroderma patients to evaluate screening tests and the incidence of pulmonary arterial hypertension and pulmonary hypertension

ELIGIBILITY:
Inclusion criteria

* Male or female
* Age ≥ 18 years
* Patients with definite diagnosis of SSc by American College of Rheumatology (ACR) criteria (18); including all patients with any other connective tissue diseases (CTD) who, in parallel, meet the ACR criteria for SSc (18)
* SSc disease duration > 3 years dated from onset of first non-Raynaud feature
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 60% of predicted

Exclusion criteria

* PH confirmed by RHC before enrolment, i.e. mean pulmonary arterial pressure (mPAP) > or = 25 mmHg at rest or > or = 30 mmHg at exercise, independent of PCWP (11)
* RHC within the 12 months before enrolment
* Use of therapy that is considered definite PAH/PH treatment (19) for any indication, within the 6 weeks before enrolment and/or for a total of more than 6 weeks during the 12 months before enrolment: i.e. endothelin receptor antagonists (ERA; e.g. bosentan, sitaxsentan, ambrisentan), phosphodiesterase type 5 inhibitors (PDE5; e.g. sildenafil, tadalafil, vardenafil), prostanoids (e.g. epoprostenol, treprostinil, iloprost, beraprost), and any experimental PAH/PH drugs. Intermittent use of PDE5 inhibitors for male erectile dysfunction is permitted
* Forced vital capacity (FVC) < 40%
* Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) < 40 ml/min/1.73 m2 (20), assessed according to local practice
* Previous evidence or previous diagnosis of clinically relevant left heart disease and other relevant conditions, i.e. at least one of the following:

  * Previous ECHO with estimated left ventricular (LV) ejection fraction < 50%, previous history of cardiogenic pulmonary edema, increased size of left atrium (> 50 mm)
  * Known significant diastolic dysfunction associated with clinical heart failure or PCWP > 15mmHg
  * Known significant coronary disease or significant valvular heart disease
  * Evidence of inadequately treated blood pressure, defined as > 160/90 mmHg and/or blood pressure during exercise > 220/120 mmHg (if evaluated)
  * Known hypertrophic cardiomyopathy or left ventricular hypertrophy (interventricular septum thickness (IVS) or posterior wall thickness (PWD) > 1.2 cm)
  * Patients referred with overt heart failure
  * Known congenital heart defects such as single ventricle, transposition, or Eisenmenger physiology
  * Previous closure of systemic pulmonary shunt, heart valve replacement, or cardiac transplantation
* Pregnancy: pregnancy testing in females with child-bearing potential is mandatory and must be done before enrolment
* Patients unlikely to be available for annual follow up over an anticipated 3 years of study (e.g. survival estimate, psychological, logistics; based on investigator discretion)

Patients with clinically relevant left heart disease as defined above, diagnosed by ECHO at baseline (i.e. after enrolment), will be included in the study.

Additional exclusion criteria after patient enrolment

* During the study, use of therapy that is considered definite PAH/PH treatment (19) is prohibited and will result in discontinuation of the patient from the study, unless the total treatment duration per year is less than 6 weeks. Intermittent use of PDE5 inhibitors for male erectile dysfunction is permitted.
* During the study, use of therapy that is considered definite PAH/PH treatment (19) is prohibited within the 6 weeks preceding the follow-up visits. Violation of this rule will result in discontinuation of the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scleroderma in USA, Canada, UK, Germany, Switzerland, Austria, The Netherlands, Belgium, Sweden, Slovakia, and Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary arterial hypertension (PAH) confirmed by right heart catheterization (RHC) | Baseline and 3-year follow-up

SECONDARY OUTCOMES:
Pulmonary hypertension (PH) confirmed by right heart catheterization (RHC) | Baseline and 3-year follow-up

CONTACTS AND LOCATIONS:
Locations (83):
- United States (23):
  - University of Alabama at Birmingham, 311 THT, Birmingham, Alabama
  - UCLA Division of Rheumatology, Los Angeles, California
  - Harbor UCLA Medical Center, Torrance, California
  - University of CT, Farmington, Connecticut
  - Department of Rheumatology, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - Rheumatology, MC 733, The University of Illinois-Chicago, Chicago, Illinois
  - John Hopkins, Division of Rheumatology, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan Scleroderma Program, Ann Arbor, Michigan
  - Michigan State University, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Division of Rheumatology, Rochester, Minnesota
  - The Center for Rheumatology, Albany, New York
  - Division of Rheumatology and Allergy - Clinical Immunology, Lake Success, New York
  - AAIR Research Center, Rochester, New York
  - Carolina Arthritis, Wilmington, North Carolina
  - Chief of Rheumatology, Toledo, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Division of Rheumatolgoy and Immunology, Charleston, South Carolina
  - Department of Critical Care - Virginia Mason Medical Center, Seattle, Washington
  - Arthritis Northwest, Spokane, Washington
  - Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin
- Austria (4):
  - Division of Pulmonology, MEDUK, Graz
  - Universitaetsklinik fuer Dermatologie und Venerologie, Innsbruck
  - Abteilung für Dermatologie, Linz
  - Univ - Klinik fuer Innere Medizin II, Abt. fuer Kardiologie - Medizinische Universitaetsklinik Wien, Vienna
- Clinic for Heart and Rheumatic Diseases, Sarajevo, Bosnia and Herzegovina
- Brazil (8):
  - Santa Casa de BH - Departamento de Reumatologia, Belo Horizonte
  - Clinical Hospital - UNICAMP University of Campinas, Campinas
  - Clinical Hospital - Federal University of Parana State - Rheumatology and Systemic Sclerosis Department, Curitiba
  - UFRJ - Serviço de Reumatologia, Ilha Do Fundão
  - Complexo Santa Casa de POA - Hospital Santa Clara, Porto Alegre
  - Hospital São Lucas da PUCRS - Pontifícia Universidade Católica de Porto Alegre (PUCRS), Porto Alegre
  - Clinical Hospital - Medicine School of the University of Sao Paulo, São Paulo
  - Clinical Hospital - Federal University of Medicine of Sao Paulo, São Paulo
- Canada (10):
  - Faculty of Medicine, Calgary, Alberta
  - 2E4.31 Walter Mackenzie Health Sciences Center, Edmonton, Alberta
  - Regent Medical Building, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre-VG Site, Halifax, Nova Scotia
  - St. Joseph Health Care, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hospital Notre-Dame, Montreal, Quebec
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - St. Paul's (Grey Nuns) Hospital, Saskatoon, Saskatchewan
- Peking Union Medical College Hospital (West Campus) Chinese Academy of Medical Sciences, Beijing, China
- Revmatologicky ustav, Prague, Czechia
- Germany (14):
  - Kerckhoff-Klinik GmbH - Abteilung Rheumatologie und Kliniscihe Immunologie, Bad Nauheim
  - Universitaetsmedizine Charite, Berlin
  - Universitaetsklinikum Bonnn, Bonn
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Medizinische Klinik 3, Rheumatologie, Immunologie und Onkologie, Erlangen
  - Goethe-Universitaet Frankfurt, Frankfurt
  - Medizinische Klinik der Albert-Ludwigs Universitaet Freiburg, Freiburg im Breisgau
  - Universitatsklinik Greifswald - Klinik fur Innere Medizin B, Greifswald
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Medizinische Klinik und Poliklinik B, Rheumatologisch Immunologische Ambulanz, Münster
  - Brüder Krankenhaus, Trier
  - University Hospital Zurich, Zurich
- Hungary (2):
  - Kardiovaszkuláris Ambulancia Kft., Debrecen
  - Pécs
- UMC St Radboud, Nijmegen, Netherlands
- Norway (3):
  - Helse Bergen HF Haukeland Universitetssykehus, Bergen
  - Rikshospitalet, University hospital of Oslo - Rheumatology department, Oslo
  - St. Olav University Hospital - Rheumatologisk avdeling, Trondheim
- Prywatny Specjalistyczny Gabinet Profesora Stanislawa, Bialystok, Poland
- UPR - Medical Sciences Campus, San Juan, Puerto Rico
- Clinica de Reumatologie, Cluj-Napoca, Romania
- State Institution "Institute of the Rheumatology of the Russian Academy of Medical Sciences", Moscow, Russia
- The National Institute of Rheumatic Diseases, Piešťany, Slovakia
- Spain (3):
  - HOSPITAL SANTA CREU i SANT PAU, Barcelona
  - Servicio de Medicina Interna Planta 2ºB, Bizkaia
  - Jefe de Servicio - Servicio de Rheumatología, Valencia
- Hopitaux Universitaires de Geneve, Geneva, Switzerland
- Turkey (Türkiye) (5):
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Adana
  - Ankara Numune Egitim ve Arastirma hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Ege Universitesi, Izmir
- Royal Free Hospital NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Gopal DM, Doldt B, Finch K, Simms RW, Farber HW, Gokce N. Relation of novel echocardiographic measures to invasive hemodynamic assessment in scleroderma-associated pulmonary arterial hypertension. Arthritis Care Res (Hoboken). 2014 Sep;66(9):1386-94. doi: 10.1002/acr.22307. PMID 24515598